CLINICAL TRIAL: NCT06683703
Title: Phase II Clinical Trial on the Efficacy and Safety of Utidelone Combined with Bevacizumab in Patients with Non-small Cell Lung Cancer with Brain Metastases.
Brief Title: Utidelone Injection Combined with Bevacizumab Injection for Non-small Cell Lung Cancer Patients with Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BG01-2401
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer Patients with Brain Metastases
Keywords: efficacy and safety
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stage 1 Safety run-in (Experimental): Utidelone + Bevacizumab
  Interventions: Drug: Utidelone combined with Bevacizumab
- Stage 1 Extension: Monotherapy group (Experimental): Utidelone
  Interventions: Drug: Utidelone
- Stage 1 Extension: Combined treatment group (Experimental): Utidelone+ Bevacizumab
  Interventions: Drug: Utidelone combined with Bevacizumab
- Stage 2 (Experimental): Utidelone + Bevacizumab
  Interventions: Drug: Utidelone combined with Bevacizumab

INTERVENTIONS:
Drug: Utidelone combined with Bevacizumab — The initial dose was Utidelone 30mg/m2/d,D1-D5,Q3W+ Bevacizumab 15mg/kg/Q3w. If dose adjustment was required due to DLT events, Utidelone was reduced by up to one dose (to 25mg/m2/d), while the dose of Bevacizumab remained unchanged (15mg/kg).
  Arms: Stage 1 Safety run-in
Drug: Utidelone — Utidelone injection, 30mg/m2/d, D1-D5 for 5 consecutive days, every 21 days as a treatment cycle
  Arms: Stage 1 Extension: Monotherapy group
Drug: Utidelone combined with Bevacizumab — In the combination group, the dose of Utidelone was determined according to the safety run-in period, 30 mg/m2/d or 25mg/m2/d, D1-D5,Q3W; The dose of Bevacizumab was 15 mg/kg/3W.
  Arms: Stage 1 Extension: Combined treatment group
Drug: Utidelone combined with Bevacizumab — The dose of Utidelone was 30 mg/m2/d or 25mg/m2/d, D1-D5,Q3W; The dose of Bevacizumab was 15 mg/kg/3w.
  Arms: Stage 2

SUMMARY:
This study is a prospective, multicenter, two-stage phase II clinical trial evaluating the efficacy and safety of Utidelone combined with Bevacizumab in patients with non-small cell lung cancer with brain metastases.

The main objective of the first stage was to determine the combined dose of the first stage and the second stage, and to compare the intracranial efficacy of the two treatment groups. Secondary objectives were to compare other intracranial efficacy, systemic efficacy, safety and tolerability between the two treatment groups.In the second stage, the main purpose was to evaluate the intracranial efficacy of Utidelone combined with Bevacizumab in patients, and the secondary purpose was to evaluate the other intracranial efficacy, systemic efficacy, safety and tolerability of Utidelone combined with Bevacizumab in patients, and to explore the improvement of patients' quality of life.

DETAILED DESCRIPTION:
Patients with non-small cell lung cancer and brain metastases were enrolled in this study. The first stage consisted of a safety run-in (combination group only) and an expansion. During the safety run-in phase, a 3+3 dose step-down design was used, starting with 30mg/m2/d of Utidelone,D1-D5,Q3W plus Bevacizumab 15mg/kg/Q3w. The dose of Utidelone was reduced by up to one dose (to 25mg per square meter), and the dose of Bevacizumab was unchanged (15mg/kg/Q3w). We planned to enroll 3 to 12 patients in the safety run-in. In the extension, the patients were randomly assigned to the combination group and the monotherapy group (hereinafter referred to as the monotherapy group). 30 patients were planned to be enrolled in the monotherapy group, and 24 or 27 patients were enrolled in the combination group according to the safety run-in. The second stage of dosing was the same as the first stage of expansion in the combination-therapy group, and the results of the first stage determined whether to proceed to the second stage. If second stage was reached, an additional 52 patients would be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent for the study was obtained from the participants and a written informed consent form (ICF) was provided.
2. age ≥18 years old and ≤70 years old, regardless of gender;
3. non-squamous non-small cell lung cancer (adenocarcinoma or adenocarcinoma component dominant) with brain parenchymal metastasis confirmed by histology or cytology, but unsuitable or refused local treatment/surgery;
4. at least one measurable intracranial lesion according to RECIST v1.1 criteria (a lesion previously treated with radiotherapy could not be considered a target lesion unless it had definite progression after radiotherapy);
5. stable brain metastases requiring no immediate or planned local treatment for brain metastases during the study;
6. driver gene negative patients, unable to tolerate standard treatment or disease progression during or after first-line treatment with platinum-based chemotherapy and immunotherapy concurrent or sequential treatment, and with brain metastasis (regardless of whether the brain metastasis had been systematically treated); Note: (new) no progression within 6 months after the last dose of adjuvant therapy does not count as line count.
7. ECOG 0-1, life expectancy > 12 weeks;
8. Patients should have adequate bone marrow reserve and no liver, kidney, or coagulation disorders. The following laboratory values should be met during screening and at baseline of enrollment:

1) Bone marrow reserve function: absolute neutrophil count ≥1.5×109/L and white blood cell count ≥3×109/L; Platelet count ≥100×109/L; Hemoglobin

* 90g/L; No blood transfusion or treatment with growth factors such as erythropoietin, thrombopoietin, or granulocyte colony-stimulating factor within 14 days; 2) Renal function: serum creatinine ≤1.5× upper limit of normal value (ULN) and creatinine clearance ≥50 mL/min (calculated according to Cockcroft and Gault formula); Urine protein <2+ (24-hour urine protein quantification within 7 days if baseline urine protein ≥2+, eligible if urine protein ≤1g) 3) Liver function: if there is no confirmed liver metastasis, AST and ALT should be ≤3×ULN; AST, ALT≤5×ULN if liver metastasis was confirmed; If there is no confirmed liver metastasis, the total bilirubin should be ≤1.5×ULN; Patients with confirmed liver metastasis or Gilbert's syndrome (indirect hyperbilirubinemia, total bilirubin ≤3×ULN); 4) Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial prothrombin time (APTT) ≤1.5×ULN. (9) Eligible patients (men and women) of childbearing potential had to agree to use a reliable contraceptive method (hormonal or barrier methods or abstinence) with their partner during the trial and for at least 3 months after the last dose; Female patients of reproductive age had to have a negative blood or urine pregnancy test before enrollment.

Exclusion Criteria:

1. primary malignant brain tumors and symptomatic or investigator-judged unstable brain metastases; Patients with leptomeningeal metastasis;
2. mixed adenosquamous carcinoma with squamous cells as the main component confirmed by histology or cytology (squamous cell carcinoma cells accounted for ≥10%);
3. The presence of EGFR, ALK, ROS1, NTRK and MET driver genes in patients with previous pathology can be determined according to the results of gene detection during the first-line treatment.
4. Patients without disease progression after whole brain radiotherapy or stereotactic conformal radiotherapy for all intracranial lesions were not eligible for measurable lesions;
5. third-space effusion (such as massive pericardial, pleural or peritoneal effusion) that could not be controlled by drainage or other methods within 4 weeks before enrollment;
6. patients received palliative radiotherapy for non-target lesions for symptom relief (e.g., pain relief by radiotherapy for bone lesions) within 2 weeks before enrollment; Patients with previous whole brain radiotherapy (WBRT) were eligible if they had received previous stereotactic radiotherapy (SRT) or other local CNS treatments (such as intrathecal chemotherapy) more than 2 weeks after the first study dose.
7. Systemic therapy: all patients had received previous anti-angiogenic drugs (bevacizumab, recombinant human endostatin, anlotinib), including previous anti-angiogenic drugs; Patients received systemic anti-tumor therapy such as chemotherapy and immunotherapy within 4 weeks before the first study medication. Traditional Chinese medicine (including patent Chinese medicine) which had received small molecule targeted therapy or tumor indication within 2 weeks before the first study medication.
8. known contraindications to gadolinium-based MRI, such as cardiac pacemaker, shraphings, or eye foreign bodies;
9. two or more seizures within 4 weeks before enrollment;
10. known to be allergic to eutideron injection, bevacizumab or any of its excipients;
11. patients with grade ≥2 peripheral neuropathy or skin abnormalities requiring treatment, or any toxicity caused by previous antineoplastic therapy that has not recovered to CTCAE grade 5.0 ≤1 (excluding grade 2 alopecia) before the first dose of the study drug;
12. There are contraindications to bevacizumab use, including but not limited to the following: - Uncontrolled severe hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥100 mmHg) - cerebral hemorrhage, These included brain metastases related to cancer - history of severe proteinuria (e.g., urine dipsticule ≥ 2+ or 24-hour urinary protein ≥ 2 g) - previous history of hypertensive crisis or hypertensive encephalopathy - history of central nervous system disease unrelated to cancer (e.g., convulsions) - vascular disease (e.g., aneurysm requiring treatment) within 6 months before the first dose of treatment. - history of hemoptysis (2 tablespoons of bright red blood per dose) within 3 months before the first dose - history of bleeding disorder or coagulation disorder in the absence of therapeutic anticoagulants - tumor involving large vessels - history of gastrointestinal perforation or fistula within 6 months before the first dose;
13. Patients with malignant tumors other than the primary tumor within 5 years before screening (cured cervical carcinoma in situ, skin basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, breast ductal carcinoma in situ, and thyroid papillary carcinoma were excluded).
14. had undergone major surgery within 4 weeks before the first dose of study medication or had not fully recovered from any previous invasive procedure;
15. use of aspirin (>325mg/ day), clopidogrel, ticlopidine, cilostazol, or other drugs known to inhibit platelet function and/or a full-dose anticoagulant within 10 days before the first dose of study medication;
16. patients with active hepatitis B and/or hepatitis C, that is, HBsAg positive and/or HBcAb positive simultaneously detected HBV DNA positive and/or anti-HCV positive and HCV RNA positive; Human immunodeficiency virus (HIV) antibody was positive; Treponema pallidum specific antibody was positive.
17. Major cardiovascular and cerebrovascular diseases occurred within 6 months before the first study medication, such as congestive heart failure (New York Heart Association functional class ≥2), acute myocardial infarction, unstable angina, QTcF > 450 ms in men or QTcF > 470 ms in women (formula: See Appendix VII), stroke, transient ischemic attack, unstable deep-vein thrombosis, arterial thrombosis, and pulmonary embolism requiring medical intervention (except infusion-related thrombosis);
18. Active infection requiring systemic therapy within 2 weeks before enrollment, such as severe pneumonia, bacteremia, sepsis, etc.; .
19. Systemic glucocorticoid therapy (more than 4 mg of dexamethasone or equivalent per day for > 3 consecutive days) within 14 days before the first study dose or planned during the study period; Patients with chronic diseases such as severe radiation pneumonitis or severe interstitial pneumonitis were treated with immunosuppressive therapy.
20. pregnant or lactating women;
21. patients who participated in other anti-tumor clinical trials and received corresponding treatment within 4 weeks before the first study medication.
22. Other reasons for not participating in the study as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial objective response rate (iORR) according to the RECIST 1.1. | Time Frame: 18 months
  iORR is defined as the proportion of subjects with a confirmed intracranial response of complete response (CR) and partial response (PR).
Determining the Expansion Dose | 18 months
  The first safety run-in phase was used to determine the dose to be administered in the combination group in the extension phase.

SECONDARY OUTCOMES:
Intracranial progression-free survival (iPFS) | Time Frame: 18 months
  iPFS: defined as time from dose index to intracranial disease progression or death from any cause.
Intracranial disease control rate (iDCR) according to the RECIST 1.1. | Time Frame: 18 months
  iDCR: defined as the proportion of subjects with confirmed intracranial response with CR, PR, and SD.
Objective Response Rate （ORR）according to the RECIST 1.1. | Time Frame: 18 months
  ORR: defined as the proportion of subjects with a confirmed CR and PR.
Disease Control Rate （DCR）according to the RECIST 1.1. | Time Frame: 18 months
  DCR: defined as the proportion of subjects with confirmed CR and PR and SD.
Progression-Free Survival, PFS | Time Frame: 18 months
  PFS : defined as time from first dose to tumor-assessed disease progression (intracranial or extracranial) or death from any cause.
Overall survival (OS) in all participants | Time Frame: Up to 2 years
  OS : defined as time from first dose to death from any cause.
Treatment-related Adverse Event-TRAE | Time Frame: Until 28 days after the last dose of treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

IPD SHARING:
Plan to Share IPD: No